CLINICAL TRIAL: NCT03418441
Title: Danish Study Group of Infections of the Brain: A Nationwide Prospective Observational Cohort Study of All Central Nervous System Infections in Adults at Departments of Infectious Diseases in Denmark
Brief Title: Central Nervous System Infections in Denmark
Acronym: DASGIB
Status: Recruiting | Type: Observational
Sponsor: Aalborg University Hospital (Other)
Collaborators: Danish Study Group of Infections of the Brain (Other)
Responsible Party: Principal Investigator, Jacob Bodilsen, Doctor, Aalborg University Hospital
Other Study IDs: DASGIB
Record Dates: First submitted 2018-01-12; First posted 2018-02-01 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Central Nervous System Infections; Bacterial Meningitis; Viral Meningitis; Aseptic Meningitis; Encephalitis; Brain Abscess; Neuroborreliosis; Neurosyphilis; Lyme Disease; Tertiary Syphilis; Cerebral Abscess; Meningitis
Keywords: Nationwide prospective observational cohort study; Epidemiology; Central Nervous System Infections; Meningitis; Encephalitis; Brain abscess; Lyme disease; Neuroborreliosis; Neurosyphilis; Tertiary syphilis
MeSH Terms: conditions — Central Nervous System Infections; Meningitis, Bacterial; Meningitis, Viral; Meningitis, Aseptic; Encephalitis; Brain Abscess; Neurosyphilis; Lyme Disease; Syphilis, tertiary; Meningitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and CSF samples are stored whenever available
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Community-acquired CNS infections — Prospective observational registration of clinical characteristics and outcome
  Other Names: bacterial meningitis; viral meningitis; encephalitis; brain abscess; neuroborreliosis; neurosyphilis

SUMMARY:
The Danish Study Group of Infections of the Brain is a collaboration between all departments of infectious diseases in Denmark. The investigators aim to monitor epidemiological trends in central nervous system (CNS) infections by a prospective registration of clinical characteristics and outcome of all adult (>17 years of age) patients with community-acquired CNS infections diagnosed and/or treated at departments of infectious diseases in Denmark since 1st of January 2015.

DETAILED DESCRIPTION:
The investigators include data on diagnosis at admission, symptoms and signs on admission, character and timing of diagnostic work-up and treatment and outcome assessed by the Glasgow Outcome Score (GOS).

Diagnostic work-up and treatment is left at the discretion of the local physician and therefore not standardised

In general any symptoms/deficits should only be listed if they are 'new' to the patient, e.g. a known palsy of the facial nerve should not be listed as a new relevant finding at admission. On the other hand, worsening of a known neurological deficit should be listed under signs in the given instrument (bacterial meningitis, encephalitis, neuroborreliosis etc). Likewise, for outcome only changes in pre-morbid conditions should be listed including place of residence, functional status, neurological deficits etc.

Time of admission is obtained in prioritized order from the ambulance charts or notifications of arrival by secretaries or nurses in the emergency departments. Timing of lumbar puncture and cranial imaging is extracted from the electronic records at the departments of biochemistry or radiology while timing of antibiotic therapy for meningitis is identified in electronic medication systems. Time to lumbar puncture, cranial imaging and antibiotic therapy is calculated as time from arrival at hospital to each of the above events.

Quality control of case enrollment is ensured by ad hoc case-to-case discussions and at study group meetings 2-3 times a year

To ensure completeness of reported CNS infections annual searches of selected International Classification of Diseases version 10 (ICD-10) codes are performed in local administrative databases at each department:

A17 A32.1 A32.7 A39.0 A52.1-52.3 A69.2 (neuroborreliosis) A83 A84 A85 A87 A89 B00.3-00.4 B01.0-01.1 B02.0-02.0 B582 B451 B375 G00 G01 G02 G03 G04 G05 G06 G07

ELIGIBILITY:
Definitions of central nervous system infections:

For all cases with unproven aetiologies no alternative diagnosis than CNS infection is thought more likely after completed multidisciplinary diagnostic work-up.

Viral meningitis inclusion criteria

- All patients have to have a clinical presentation consistent with non-bacterial meningitis (e.g. headache, neck stiffness, photo- or phonophobia, fever)

and

Cerebrospinal fluid leukocytes>10 cells/ml

Patients with viral meningitis with undetermined pathogen have to have:

* CSF leukocytes> 10/mL and no other more probable diagnosis assessed by the local investigator.

In case of doubt, patients are discussed with the DASGIB secretary and chair or at meetings.

Bacterial meningitis inclusion criteria - All patients have to have a clinical presentation consistent with bacterial meningitis (e.g. headache, neck stiffness, fever, altered mental status)

and

Proven bacterial aetiology (CSF or blood culture/DNA based technology or antigen tests)

Patients with bacterial meningitis in whom the bacteria cannot not be cultured or identified by DNA-based technologies have to have:

- CSF leukocytes> 10/mL and no other more probable diagnosis assessed by the local investigator.

In case of doubt, patients are discussed with the DASGIB secretary and chair or at meetings.

Encephalitis inclusion criteria - All patients have to have a clinical presentation consistent with encephalitis (e.g. headache, fever, focal neurological deficit, altered mental status >24 hours) as defined by the International Encephalitis Consortium (Venkatesan A et al., Clin Infect Dis 2013; doi:10.1093/cid/cit458.).

Encephalitis exclusion criteria

- We exclude cases of proven or suspected autoimmune encephalitis.

Primary brain abscess inclusion criteria

- All patient have a clinical presentation consistent with brain abscess (e.g. headache, focal neurological deficit, mass lesion on cranial imaging)

and

- Proven microbiological aetiology by culture/DNA-based technology from pus from brain abscess or blood or CSF

or

- Aspiration of pus from the brain abscess

or

- Response to antimicrobial treatment

or

- Tumour ruled out

or

- Tumour thought less probable than abscess on MRI using diffusion weighted imaging (DWI) and apparent diffusion coefficient (ADC) sequences.

Lyme neuroborreliosis inclusion criteria

- A clinical presentation consistent with neuroborreliosis (e.g. radiculopathy)

and

- CSF pleocytosis>10 leukocytes/mL

and

- Positive intrathecal B.burgdorferi antibody production index.

Neurosyphilis inclusion criteria - A clinical presentation consistent with neurosyphilis (e.g. 'encephalitis-like symptoms', dementia, ocular or otogenic syphilis)

and either

- Positive syphilis serology in serum combined with CSF leukocytes>10/mL

or

- CSF syphilis antibodies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients above 17 years of age are prospectively included in the DASGIB cohort by the principal investigator at each site if they have a clinical presentation suggestive of CNS infection (e.g. any combination of neck stiffness, fever, headache or altered mental status) and either (i) Positive CSF culture or positive bacterial/viral DNA-based analysis for (community-acquired) pathogens in the CSF or (ii) a positive blood culture and CSF leukocytes >10/mL or (iii) CSF leukocytes > 10/mL without any alternative diagnoses more likely to explain the patients' conditions. Exceptions apply for brain abscess, neurosyphilis and neuroborreliosis and exact definitions of included CNS infections are provided below.
  We exclude patients with hospital-acquired CNS infections as defined by the Centers for Disease Control and Prevention (Garner et al, Am J Infect Control, 1988), or an implanted neurosurgical device.
Sampling Method: Non-Probability Sample
Enrollment: 1900 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2030-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Incidence | One year
  Incidence of CNS infections in the adult population (>17 years of age) in Denmark.

SECONDARY OUTCOMES:
Glasgow Outcome Scale score | One month after end of treatment
  A five tier assessment of functional status, 1=Death, 2=vegetative state, 3=dependency on others for daily activities, 4=some sequelae but able to live independently, 5= No or only minor sequelae
Glasgow Outcome Scale score for viral meningitis | 30 days
  A five tier assessment of functional status, 1=Death, 2=vegetative state, 3=dependency on others for daily activities, 4=some sequelae but able to live independently, 5= No or only minor sequelae
Glasgow Outcome Scale score for bacterial meningitis | 30 days
  A five tier assessment of functional status, 1=Death, 2=vegetative state, 3=dependency on others for daily activities, 4=some sequelae but able to live independently, 5= No or only minor sequelae
Glasgow Outcome Scale score for encephalitis | 30 days
  A five tier assessment of functional status, 1=Death, 2=vegetative state, 3=dependency on others for daily activities, 4=some sequelae but able to live independently, 5= No or only minor sequelae
Glasgow Outcome Scale score for neurosyphilis | 2 weeks
  A five tier assessment of functional status, 1=Death, 2=vegetative state, 3=dependency on others for daily activities, 4=some sequelae but able to live independently, 5= No or only minor sequelae
Glasgow Outcome Scale score for neuroborreliosis | 2 weeks
  A five tier assessment of functional status, 1=Death, 2=vegetative state, 3=dependency on others for daily activities, 4=some sequelae but able to live independently, 5= No or only minor sequelae
Glasgow Outcome Scale score for brain abscess | 8 weeks
  A five tier assessment of functional status, 1=Death, 2=vegetative state, 3=dependency on others for daily activities, 4=some sequelae but able to live independently, 5= No or only minor sequelae

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Nielsen, Professor, Study Chair — Aalborg University Hospital
Locations (8):
- Denmark (8):
  - Department of Infectious Diseases, Aalborg University Hospital, Aalborg
  - Department of Infectious Diseases, Aarhus University Hospital Skejby, Aarhus
  - Department of Infectious Diseases, Rigshospitalet, Copenhagen
  - Herlev-Gentofte Hospital, Copenhagen
  - Department of Pulmonary and Infectious Diseases, Nordsjællands Hospital Hillerød, Hillerød
  - Department of Infectious Diseases, Hvidovre Hospital, Hvidovre
  - Department of Infectious Diseases, Odense University Hospital, Odense
  - Department of Pulmonary and Infectious Diseases, Sjællands University Hospital Roskilde, Roskilde

IPD SHARING:
Plan to Share IPD: Undecided